CLINICAL TRIAL: NCT00749489
Title: Improving Pain and Function in Hip Fracture
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 06-0721; AG030141-01 A1 (Other Grant/Funding Number: National Institute on Aging (NIA))
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Pain; Hip Fractures
Keywords: Pain; Hip Fractures; Femoral Fractures; Analgesics; Opioid; Nerve Block; Geriatric; Nerve Stimulation
MeSH Terms: conditions — Pain; Hip Fractures; Femoral Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Femoral Nerve Block (Experimental): Intervention patients will have a continuous fascia iliaca blocks placed by a regional anesthesiologist 24 hours after the initial single injection femoral nerve block or at the time of surgery.
  Interventions: Procedure: Femoral Nerve Block
- No Intervention (No Intervention): No intervention

INTERVENTIONS:
Procedure: Femoral Nerve Block — Patients assigned to the intervention group will have a femoral nerve block administered by the attending emergency department physician. Twenty-four hours after the femoral nerve block or at the time of surgery, an anesthesiologist will insert a continuous fascia iliaca block. Both procedures (femoral nerve block and fascia iliaca blocks) are standard anesthetic techniques that are used in orthopedic procedures but their efficacy as compared to standard opioid therapy has not been evaluated in controlled clinical trials in hip fracture. The medications that will be used in each procedure are as follows: 1) femoral nerve block: 0.5% bupivacaine with 1:300,000 epinephrine; 2) fascia iliaca block: 0.2% ropivacaine will be infused at 5ml/hr.
  Arms: Femoral Nerve Block

SUMMARY:
The purpose of this study is to compare two different methods of treating pain after a hip fracture.

DETAILED DESCRIPTION:
This project examines the efficacy and effects of 2 regional anesthesia techniques, femoral nerve blocks (FNB) and fascia iliaca blocks (FIB), on the treatment of peri-operative acute hip (femoral neck, intertrochanteric) fracture pain. Patients age 60 years and over presenting to two New York City emergency departments with hip fracture will be randomized to receive the intervention or usual care. The intervention includes single injection FNB in the ED followed by insertion of a continuous FIB catheter within 24 hours of the single injection FNB plus "as needed" non-opioid/opioid analgesia. Usual care patients will receive conventional therapy with regularly scheduled intravenous or oral opioids plus "as needed" non/opioids/opioids. We will examine the impact of the intervention on patients' self reported pain intensity; systemic opioid requirements; post-operative function; incidence of delirium, treatment related side effects; and hospital length of stay and participation in physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients 60 years of age and over that present to the MSMC ED from 8:00 to 20:00 with a radiographically confirmed hip fracture (femoral neck, intertrochanteric, or peri-capsular) will be screened for study eligibility.

Exclusion Criteria:

* History of advanced dementia
* Presence of multiple trauma, pathological fractures, bilateral hip fractures, or previous fracture or surgery at the currently fractured site
* Patients transferred from another hospital
* Patients with cirrhosis or liver failure.
* The investigators exclude patients with advanced dementia because the investigators will require patients to self-report their pain intensity.
* The investigators exclude these categories of hip fracture because they represent patients with atypical or often problematic clinical circumstances.
* The investigators exclude patients under age 60 because our focus is on treatment of pain in older adults. Younger adults (less than age 60) typically present with fractures of different cause (severe and multiple trauma), are less sensitive to the side effects and complications of opioid therapy, are less likely to have delayed or prolonged functional recovery, and are less sensitive to the adverse and sometimes permanent effects of prolonged bed rest (i.e., from pain) on function.
* The investigators exclude patients with hepatic dysfunction because the intervention protocol includes administration of acetaminophen which can provoke liver failure in patients with advanced liver disease.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2008-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pain; 11-point Numeric Rating Scale | three times daily for pain for the duration of hospital stay (average stay is 4 days)

SECONDARY OUTCOMES:
Delirium; Confusion Assessment Method (CAM). | three times daily for pain for the duration of hospital stay (average stay is 4 days)

CONTACTS AND LOCATIONS:
Overall Officials: R. Sean Morrison, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Knox Todd, MD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Beth Israel, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Maimonides Medical Center, New York, New York

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043
- See also: National Palliative Care Research Center — http://www.npcrc.org